CLINICAL TRIAL: NCT03602183
Title: A Comparison of Direct vs. Video-laryngoscopes for Different Emergency Pediatric Airway Scenarios
Brief Title: Pediatric Intubation During Emergency Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Collaborators: Wroclaw Medical University (Other); The Cleveland Clinic (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Associate Professor, Lazarski University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI_2018_PALS
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Endotracheal Intubation; Pediatric; Cardiac Arrest; Injuries
Keywords: difficult airway; endotracheal intubation; chest compression; physician
MeSH Terms: conditions — Heart Arrest; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal airway scenario (Experimental): intubation in normal airway scenario
  Interventions: Device: Macintosh laryngoscope; Device: Miller laryngoscope; Device: McGrath MAC EMS; Device: GlideScope
- Tongue edema scenario (Experimental): intubation in the tongue edema scenario. Tongue edema was obtain using simulator indicators
  Interventions: Device: Macintosh laryngoscope; Device: Miller laryngoscope; Device: McGrath MAC EMS; Device: GlideScope
- Spinal immobilization with normal airway scenario (Experimental): intubation in spinal immobilization with normal airway scenario
  Interventions: Device: Macintosh laryngoscope; Device: Miller laryngoscope; Device: McGrath MAC EMS; Device: GlideScope
- Spinal immobilization with tongue edema scenario (Experimental): endotracheal intubation with immobilized cervical spine and tongue edema scenario
  Interventions: Device: Macintosh laryngoscope; Device: Miller laryngoscope; Device: McGrath MAC EMS; Device: GlideScope

INTERVENTIONS:
Device: Macintosh laryngoscope — intubation will be performed using standard direct laryngoscopy - Macintosh laryngoscope
  Other Names: MAC
Device: Miller laryngoscope — intubation will be performed using Miller laryngoscope
  Other Names: MIL
Device: McGrath MAC EMS — intubation will be performed using McGrath MAC EMS video - laryngoscope
  Other Names: McGrath
Device: GlideScope — intubation will be performed using GlideScope video - laryngoscope
  Other Names: GLS

SUMMARY:
The effectiveness of endotracheal intubation in pre-hospital conditions is insufficient - especially in the context of pediatric patients. Anatomical differences in pediatric patients compared to adults: a relative larger tongue, a larger and more flabby epiglottis - located more cephalously - that make intubation is more difficult than for adults. Also, higher oxygen metabolism requires the immediate response of medical personnel to children in case of need to protect the airways and support breath.

ELIGIBILITY:
Inclusion Criteria:

* paramedics
* give voluntary consent to participate in the study
* none experience in videolaryngoscopy
* less than 1 year experience in medicine

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Intubation time | 1 day
  time in seconds required for a successful intubation attempt

SECONDARY OUTCOMES:
Success of intubation | 1 day
  If the oesopharyngeal tube was incorrectly placed or intubation lasted longer than 60 seconds, the airway-management attempt was defined as a failure.
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading, scale developed by Cormack and Lehane, based on four degrees of visibility of the glottis.
POGO score - percentage of glottic opening | 1 day
  self-reported percentage the vocal cord visualization. A 100% POGO score is a full view of the glottis from the anterior commissure to the interarytenoid notch. A POGO score of 0 means that even the interarytenoid notch is not seen.
Preferred ETI device | 1 day
  participants were asked which method of ETI they would prefer in a real-life resuscitation.
Ease of use | 1 day
  self-reported percentage the vocal cord visualization. A 100% score is a extremely difficult procedure. A Ease of use score of 1% means that procedure is extremely easy

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, PhD, Principal Investigator — Lazarski University
Locations (1):
- Lazarsku University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
data will be available from the main investigator

REFERENCES:
- [Background] Szarpak L, Karczewska K, Czyzewski L, Truszewski Z, Kurowski A. Airtraq Laryngoscope Versus the Conventional Macintosh Laryngoscope During Pediatric Intubation Performed by Nurses: A Randomized Crossover Manikin Study With Three Airway Scenarios. Pediatr Emerg Care. 2017 Nov;33(11):735-739. doi: 10.1097/PEC.0000000000000741. PMID 27228145
- [Background] Madziala M, Smereka J, Dabrowski M, Leung S, Ruetzler K, Szarpak L. A comparison of McGrath MAC(R) and standard direct laryngoscopy in simulated immobilized cervical spine pediatric intubation: a manikin study. Eur J Pediatr. 2017 Jun;176(6):779-786. doi: 10.1007/s00431-017-2909-9. Epub 2017 Apr 21. PMID 28429117
- [Background] Szarpak L, Kurowski A, Czyzewski L, Rodriguez-Nunez A. Video rigid flexing laryngoscope (RIFL) vs Miller laryngoscope for tracheal intubation during pediatric resuscitation by paramedics: a simulation study. Am J Emerg Med. 2015 Aug;33(8):1019-24. doi: 10.1016/j.ajem.2015.04.054. Epub 2015 Apr 30. PMID 25979300